CLINICAL TRIAL: NCT06533761
Title: A Phase 1b Open-Label Study to Evaluate the Safety and Tolerability of Eganelisib as Monotherapy and in Combination With Cytarabine in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Eganelisib as Monotherapy and in Combination With Cytarabine in Relapsed/Refractory AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stelexis BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STLX-EGA-001
Record Dates: First submitted 2024-07-24; First posted 2024-08-01 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: AML, Adult; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eganelisib (Experimental)
  Interventions: Drug: Eganelisib
- Eganelisib in combination with cytarabine (Experimental)
  Interventions: Drug: Eganelisib in combination with cytarabine

INTERVENTIONS:
Drug: Eganelisib — eganelisib will be administered as monotherapy
  Arms: Eganelisib
Drug: Eganelisib in combination with cytarabine — eganelisib will be administered in combination with cytarabine
  Arms: Eganelisib in combination with cytarabine

SUMMARY:
This is a Phase 1b open-label, multicenter, dose-escalation and dose-optimization study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and anti-tumor efficacy of eganelisib as monotherapy and in combination with cytarabine in patients with relapsed/refractory (r/r) acute myeloid leukemia (AML) or r/r higher-risk myelodysplastic syndromes (HR-MDS).

The study consists of 2 parts:

* Part 1: Dose Escalation (DE) in both monotherapy and in combination.
* Part 2: Dose Optimization

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of either: AML according to World Health Organization (WHO) 2022 revised criteria per the local pathology report and with ≥10% bone marrow blasts (acute promyelocytic leukemia is excluded but secondary AML and treatment-related AML can be included); Higher-risk (IPSS-R Intermediate, High or Very High Risk at time of study entry) myelodysplastic syndromes (HR-MDS) according to WHO 2022 revised criteria per the local pathology report and with ≥10% bone marrow blasts.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Adequate hepatic and renal function measured within 7 days prior to the first dose of eganelisib.

Exclusion Criteria:

* Autologous or allogeneic stem cell transplant within 6 months prior to Cycle 1 Day 1.
* Receiving immunosuppressants (eg, cyclosporin) or systemic steroids (except for steroid use as cortisol replacement therapy in documented adrenal insufficiency).
* Active fungal disease or uncontrolled infection of any kind; patients receiving antibiotic, antifungal or antiviral treatment must be afebrile and hemodynamically stable for >72 hours prior to treatment
* WBC count >25 × 10^9/L measured within 7 days prior to the first dose of eganelisib (hydroxyurea is permitted to decrease the WBC count).
* Presence of a clinically significant non-hematologic toxicity of prior therapy that has not resolved to Grade ≤1 or Baseline, whichever is worst, as determined by NCI CTCAE v 5.0, except alopecia or skin pigmentation. Fatigue and neuropathy must have resolved to Grade ≤2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs), graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0 | 12 months
Incidence and severity of dose-limiting toxicities (DLTs) in DLT evaluable patients during Cycle 1 | 28-35 days
Preliminary clinical activity as evaluated per European LeukemiaNet (ELN) 2022 criteria for AML and International Working Group (IWG) 2023 criteria for HR-MDS | 12 months

SECONDARY OUTCOMES:
Area under the plasma concentration time curve extrapolated to the last measurable time point [AUClast] of eganelisib and cytarabine | 112 days
Maximum concentration [Cmax] of eganelisib and cytarabine | 112 days
Time of maximum concentration [Tmax] of eganelisib and cytarabine | 112 days
Plasma half-life [t1/2] of eganelisib and cytarabine | 112 days
Measure plasma concentrations of eganelisib and determine model-based PK parameters | 112 days

CONTACTS AND LOCATIONS:
Locations (12):
- United States (10):
  - City of Hope, Duarte, California
  - Anshutz Cancer Pavilion, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University in St Louis, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
- Spain (2):
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No